CLINICAL TRIAL: NCT06700772
Title: Histomorphometric and Radiographic Assessment of Bone Following Maxillary Sinus Augmentation Using Bone Marrow Concentrate Cells From the Maxillary Tuberosity Mixed With Bovine Bone Versus Autogenous Bone Mixed With Bovine Bone: RCT
Brief Title: Histomorphometric and Radiographic Evaluation of Bone Following Maxillary Sinus Augmentation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Megahed Hassan Abdullah, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-12-5-2024
Record Dates: First submitted 2024-11-16; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Sinus Floor Elevation
Keywords: Bone replacement materials; Bone substitutes; Maxillary sinus augmentation

STUDY DESIGN:
Intervention Model Description: A Randomized clinical trial A trial will be conducted in hospital of oral and maxillofacial surgery department.faculty of oral and dental medicine Cairo university Equal randomization of participant Both groups receiving treatment Each group of patient receiving a single treatment simultaneously
Masking Description: None. Because the two interventions used in this trial are clearly different and can be easily recognized by the participant and investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- open sinus lifting using bone marrow aspirate from maxillary tuberosity mixed with bovine bone (Experimental): Under local anesthesia a 20 gauge needle that will be inserted inside tuberosity until aspiration is positive and then the aspirate will be collected in heparin treated tube (1ml anticoagulant citrate dextrose) for each 15 ml of aspirate The aspirate will be centrifuged at 3000 rpm for 10 minutes to separate the BMAC The upper layer containing the plasma and platelet will be separated using sterile peptide tube leaving the BMAC Mixing BMAC with bovine bone (2cc of bio-oss) and it will be applied in grafted sinus
  Interventions: Procedure: mixing bone marrow aspirate concentrate from maxillary tuberosity with bovine bone
- Open sinus lifting using autogenous bone mixed with bovine bone (Active Comparator): After injection of local anesthesia a crystal incision will be done from a point corresponding to occlusal surface along external oblique ridge and extending anteriorly and inferiorly through the buccal mucosa Subperiosteal dissection will be done to expose the retromolar area ACM bur will be used to collect autogenous bone and mixing it with bovine bone 50 : 50 Then this mixture will be packed into the grafted area
  Interventions: Procedure: mixing autogenous bone with bovine bone

INTERVENTIONS:
Procedure: mixing bone marrow aspirate concentrate from maxillary tuberosity with bovine bone — open sinus lifting using bone marrow aspirate concentrate from maxillary tuberosity and mixing it with bovine bone .
  Arms: open sinus lifting using bone marrow aspirate from maxillary tuberosity mixed with bovine bone
Procedure: mixing autogenous bone with bovine bone — open sinus lifting using autogenous bone from retromolar area mixed with bovine bone
  Arms: Open sinus lifting using autogenous bone mixed with bovine bone

SUMMARY:
Two groups of patients with posterior vertical deficient maxillary alveolar ridge with pneumatized sinus and needing dental implant . First group will be subjected to open sinus lifting using autogenous bone mixed with bone marrow aspirate concentrate cells from maxillary tuberosity and the second group will be subjected to open sinus lifting using autogenous bone mixed with bovine bone

DETAILED DESCRIPTION:
Two groups of patients with partial edentulous posterior maxilla with pneumatized sinus and need dental implant. First group will be subjected to open sinus lifting using autogenous bone mixed with bone marrow aspirate concentrate cells from maxillary tuberosity (the study group) and the second group will be subjected to open sinus lifting using autogenous bone mixed with bovine bone (control group) Intervention Eligible patients will be equally randomized in a parallel two arm groups . The study group (open sinus lifting using bone marrow aspirate concentrate from maxillary tuberosity mixed with bovine bone) Procedure will be performed under local anesthesia A 20 gauge needle will be inserted in the maxillary tuberosity area through the palatal aspect until aspiration is positive.

Aspirate will be collected in a heparin-treated tube (2000:1) using 1ml of anticoagulant acid citrate dextrose solution for every 15ml of bone marrow aspiration.

Aspirate will be centrifuged at 3000 rpm for 10 minutes to separate the BMAC . The upper layer containing plasma and platelets will be collected using a sterile pipette, leaving the bone marrow aspirate bone marrow aspirate will be mixed with bovine bone and then the mixture will be applied in open sinus lifting Control group (open sinus lifting using autogenous bone from retromolar area mixed with bovine bone) After injection of local anesthesia a crestal incision will be carried out from a point corresponding to the occlusal surface along the external oblique ridge and extending anteriorly and inferiorly through the buccal mucosa, parallel to the gingival margin of the mandibular molars.

The subperiosteal dissection will be extended to expose the ascending ramus and the retromolar region.

Auto chip maker bur will be used to drill out some autogenous bone particulate from retromolar which will be mixed with xenogeneic graft with a 50% to 50% ratio respectively. this mixture will be packed into the grafted site .

Post operative instructions and follow up:

Administration of:

1. Antibiotics (Amoxicillin 1g twice daily for 5 days) to prevent any chance of infection.
2. Anti-inflammatory drugs (NSAIDS; Ibuprofen 600mg three times daily for 5 days) to avoid any chance of edema or pain or swelling
3. Antiseptic mouth rinse (0.12% Chlorhexidine oral rinse will be prescribed for 60 seconds two times a day for 14 days.

   * The patient will be instructed to follow up for the next months before implant placement

Patient self-care instructions:

1. Application of an ice bag to the treated area for the first 24 hours.
2. Avoid any brushing and trauma to the surgical site for one week
3. avoid smoking
4. The patient will be asked to keep on clear fluid diet for the first 24 hours then a soft diet to be maintained for the next day.
5. Strict oral hygiene measures in the form of regular use of toothbrush and antiseptic mouthwash starting week after surgery. Warm saline oral rinsing three times daily for one week.

Postsurgical procedure (six months lateral sinus lifting) Local anaesthesia will be administered by infiltration or nerve block to achieve the necessary anaesthesia.

A flap will be raised at the presurgical site. A core biopsy will be harvested by introducing a core drill bit in place of an initial drill.

Sequential drilling will take place to prepare osteotomy to the right size to receive an implant.

Implant will be placed in the osteotomy with the platform flush with the bone. Flap closure will be achieved by interrupted 5-0 sutures. Outcomes Primary outcome quantity of bone gain Secondary outcome quality of bone gain

ELIGIBILITY:
Inclusion Criteria:

1. Patients with missing maxillary teeth with pneumatized sinus and remaining bone height <5mm
2. Patients with healthy systemic condition (Medically free)
3. Adequate inter-arch space for placement of the implant prosthetic part.
4. Good oral hygiene
5. Cooperative patients who are willing to commit for 6 months follow up

Exclusion Criteria:

1. Smokers
2. Pregnant females
3. Patient with medical condition that contraindicates surgical procedures.
4. Patients on medication that may interfere with healing (corticosteroids, bisphosphonate, Chemo/radio therapy).
5. Patients with habits that may jeopardize the implant longevity and affect the results of the study such as alcoholism or parafunctional habits.
6. Patients have chronic sinus disease.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic assessment | 6 months postoperative
  Calculation of vertical bone gain quantity using cone beam computed tomography

SECONDARY OUTCOMES:
Histomorphometric analysis | 6 months postoperative
  Assessment of bone quality after open sinus lifting this bone will be harvested using trephine bur .and bone analysis will be done using H&E stain by microscope

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Mounir shaker, Study Director — Faculty of oral and dental medicine cairo university
Locations (2):
- Egypt (2):
  - Faculty of oral and dental medicine - cairo university, Cairo, New Cairo
  - Faculty of oral and dental medicine - cairo university, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Human maxillary tuberosity and jaw periosteum as sources of osteoprogenitor cells for tissue engineering. — https://pubmed.ncbi.nlm.nih.gov/17613258/
- See also: Stem cells in dentistry--part I: stem cell sources. — https://pubmed.ncbi.nlm.nih.gov/22796367/